CLINICAL TRIAL: NCT06337370
Title: Self-management Nursing Intervention for Women With Rheumatoid Arthritis: A Pragmatic Randomized Clinical Trial
Brief Title: Self-management Nursing Intervention for Women With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Ministerio de Ciencia Tecnología e Innovación - Minciencias (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 61284
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: Chronic disease self management program; Women; Arthrits rheumatoid; Health related quality of life; Selfmanagement; Self efficacy; Pragmatic randomized controlled trial
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: CDSMP is a group-based chronic disease self-management education intervention comprised of 2.5-hour sessions, including time for a break and snack. The maximum number of participants per session ranges from 12 to 16. In total the program consists of 6 sessions that take place once a week for a total duration of 6 weeks. The development of each of the sessions is standardized and scripted; two group leaders previously trained by a Master Trainer, who in turn was trained to train leaders with Stanford University, guide the sessions. In the case of the present study, the main researcher and a nursing professional with experience in health education will receive the training from a Master Trainer of the program. Participants receive the book "Taking Control of Your Health" at the beginning of the program.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In order to guarantee the objectivity and impartiality of the research team, randomization will be accompanied by blinding. A single-blind trial is proposed in which the participants during the conduct of the study will be unaware of their assignment to the experimental or control groups; likewise, the research assistants who perform the pre and post measurement will be unaware of their assignment to the groups; there will be specific assistants for the pre measurement and specific assistants for the post measurement with each group. Candidates will be invited to participate in the study, explaining to them that it is a randomized study in which they may be assigned to a specific intervention group, that their assignment will only be random, that neither the research team nor the treating health team will be able to interfere with their assignment and that this will be revealed to them once the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSMP Group (Experimental): Participants will receive the chronic disease selfmanagement program for 6 weeks.
  Interventions: Behavioral: Chronic Disease Self Management Program
- Conventional Care Group (Active Comparator): Participants will receive conventional care.
  Interventions: Behavioral: Conventional Intervention- Standard care

INTERVENTIONS:
Behavioral: Chronic Disease Self Management Program — Experimental Intervention (Self-Management Program):
  In addition to standard care from a rheumatology specialist, the intervention group will receive the Chronic Disease Self-Management Program (CDSMP). This program is a group intervention that provides education on self-managing chronic diseases. The program consists of six weekly sessions, each lasting two and a half hours (including time for breaks and refreshments), for a total of six weeks. Each group will consist of 12 to 16 participants, and the sessions will follow a standardized, scripted format. Two group leaders, who have received training from a Master Trainer certified by Stanford University in how to implement the program, will lead the activities. For this study, the principal investigator and a nurse experienced in health education will undergo training from a CDSMP Master Trainer to ensure fidelity to the intervention.
  Arms: CDSMP Group
Behavioral: Conventional Intervention- Standard care — Conventional intervention (standard care):
  The control group will receive standard care provided by a rheumatology specialist. This approach emphasizes clinical and clinimetric evaluations of rheumatoid arthritis. It includes applying validated disease activity indices (e.g., DAS28, CDAI, or SDAI), making therapeutic decisions, and adjusting medications according to current clinical practice guidelines. It also includes the standard clinical counseling provided during routine medical consultations. No additional self-management strategies or structured interventions beyond those already incorporated into routine healthcare practice will be included.
  Arms: Conventional Care Group

SUMMARY:
Introduction. Chronic autoimmune diseases are catalogued as catastrophic conditions that generate a negative impact on the health and well-being of the affected person. In this particular case, rheumatoid arthritis (RA) is its main representative, which is a predominant disease in women, affecting not only the musculoskeletal system but in general, all dimensions of the human being and generating great costs for health systems. Adaptation to living with the disease requires the individual to develop capacities for a positive management of the condition, and in this sense, the development of self-management behaviors becomes a crucial element. Method. The investigators propose a two-arm pragmatic randomized clinical trial with pre- and post-intervention measures, to evaluate the effect of the Chronic Disease Selfmanagement Program (CDSMP) on the increase in the levels of self-efficacy, self-management and health-related quality of life of women with RA who are attended by outpatient rheumatology consultation in a health institution in Bogota compared to usual care. Results. A description will be made of the sociodemographic and clinical variables present in you together with the measurement of the variables of health-related quality of life through the Quality Of Life-Rheumatoid Arthritis Scale-II (QOLRA-II); self-efficacy with the specific scale of self-efficacy in arthritis; and self-management behaviors by means of the scale of self-management in the disease. The measurement for the intervention group will be performed before and after the implementation of the program and for the control group an initial measurement and another one after six weeks. Discussion. The implementation of the CDSMP could generate a positive effect on the variables of self-management, self-efficacy and health-related quality of life in women with RA who are attended by outpatient consultation in a health institution in Bogota compared to usual care.

DETAILED DESCRIPTION:
Statement of the problem Inflammatory rheumatic diseases, as chronic degenerative diseases, represent a high expense for the General Social Security Health System (SGSSS) reflected in the costs of care and the affectation in the personal, labor, social and family spheres that cause a deterioration in the quality of life related to the health of the individual.

The main representative of this group is RA, considered as a chronic and disabling systemic disease affecting joints, connective tissue, muscles, tendons and fibrous tissue. By causing pain and deformity, it is one of the main causes of absenteeism and premature retirement from work in the world.

However, the general age of onset is in adulthood. In the interval between 55 and 59 years of age, about 50% of people suffering from this condition, after 10 years, have lost their ability to work or are unable to maintain a full-time job.

Looking at Colombia, figures reveal that 2.2% of the general population suffers from RA. Specifically, for the year 2022, a total of 118,497 cases were reported, of which 5,115 were incidents with a percentage increase of 41.53 % compared to the previous period and, of these, 81.52 % are women, with a female-to-male ratio of 4.41 to 1. Regarding the situation observed in Bogotá, the High-Cost Account (CAC) states that this is one of the regions with the highest number of cases reported by the territorial entities: 28,012 for the year 2022.

Because of the personal, physical, occupational, family and social impact it produces on the health and well-being of the affected population, RA is classified as a ruinous, catastrophic, progressive, high-cost disease of public health interest. Specifically, its presence in the female population represents a source of low levels of health-related quality of life (HRQoL).

In this sense, Corbin and Strauss, regarding the impact of chronic disease on patients' lives, state that their experience requires the fulfillment of three types of tasks: management of the disease seen as the clinical management of the condition, management of the role in terms of behavioral management and management of the emotions associated with the new experience. In the case of women with RA, the Pan American League of Rheumatology Associations (PANLAR) and the Latin American Group for the Study of RA (GLADAR) highlight the implementation of interventions aimed at improving self-management as one of the priorities for health care in Latin America.

According to Grady and Gough, self-management is a highly effective strategy to address chronic diseases because it offers people, in addition to information, the necessary tools to detect and solve the problems associated with their disease.

Lorig & Holman state that, because RA is a chronic condition that accompanies and modifies the patient's life from the moment of diagnosis, it requires participation focused on resolving the difficulties that the disease brings with it, managing resources and making informed decisions that allow him/her to adopt or restructure behaviors to live fully.

Currently, nursing interventions are available that have addressed self-management in chronic conditions such as RA, aimed at developing in the person the ability to self-manage their health reflected in self-management behaviors; however, the available evidence on their effect in Latin American countries has not been evaluated and the cost for their implementation and validation is very high.

In this sense, although in Latin America there are no specific self-management programs for the care of people with RA, there is a generic self-management program for chronic diseases -Chronic Disease Self Management Program- called in Spanish "Tomando el control de su salud", validated in some states of Mexico, by Peñarrieta and his research group at the Autonomous University of Tamaulipas with support from the Pan American Health Organization.

Both the specific self-management program for RA and the generic self-management program for chronic diseases were designed at Stanford University and when comparing them, the authors describe that both programs show positive results in health, that although the specific program can show advantages 4 months after the post-intervention measurement, these advantages are reduced after one year, concluding that the CDSMP program is a viable alternative when resources are not sufficient and suggesting that with the implementation of a generic program it is possible to reach a greater number of people at a lower cost, a similar situation occurred in the case of the CDSMP program, a similar situation occurred in the study by Goeppinger who, when comparing the effect of both programs in the African American population with RA, found statistically significant differences in pain and disability for both groups 4 months after implementation; in this case, the CDSMP showed better results.

The evaluation of the effect of the CDSMP program in Latin countries has only been measured in Tampico, Mexico, by Peñarrieta, who through a two-arm experimental approach: intervention group and control group applied it to patients with chronic diseases attended in first level care institutions, in their results they describe that the program is effective in improving health and self-management behaviors in adults with diabetes and arterial hypertension in Tampico, however, they highlight the need to continue conducting research to understand the effect of the self-management program in NCDs in the different regions of Mexico and the rest of Latin America, they suggest using objective measures with a longer follow-up; they state as limitations: a small sample size and the measurement of dependent and independent variables with self-report scales, increasing the possibility of bias.

To understand the mechanisms involved in the adoption of self-management behaviors, it is essential to take into account psychosocial aspects such as self-efficacy, i.e., the belief in each person's ability to organize and execute the courses of action necessary to produce certain achievements. The CDSMP program is based on Bandura's theory of self-efficacy, which identifies it as a determining factor for the adoption of health behaviors and decision making.

Thus, recognizing the negative impact and burden of rheumatoid arthritis on the health and well-being of women and the great contribution that the nursing discipline can offer through its intervention, the present research proposal is proposed as a novel approach that aims to evaluate the effect of a self-management intervention - CDSMP - for women with RA in Bogota.

Study Justification The nursing intervention in self-management for women with RA finds its justification in the chronic condition of the disease that implies that people play an active role in the control of their symptoms, in the anticipation of complications and in the possibility of being managers of health behaviors in benefit of their health-related quality of life. For such reason, there is a growing need to evidence the effect of nursing interventions in self-management on chronic disabling conditions, such as RA in Latin America.

This research, therefore, proposes an innovation in nursing care for the health of women with RA, which corresponds to the integration of a self-management intervention with empirical support and the consideration of psychosocial variables such as self-efficacy and health-related quality of life. This is intended to help reduce the disarticulation that exists between the welfare approach and the Primary Health Care (PHC) approach, which transcends the consideration of people's particularities. Likewise, the self-management and self-efficacy behaviors that could generate benefits in health-related quality of life will be known in greater depth.

Research Question Is the self-management intervention - CDSMP - effective in increasing levels of self-efficacy, self-management behaviors and health-related quality of life (HRQOL) of women with RA seen in outpatient care at a health institution in Bogota compared to conventional care?

General Objective To evaluate the effect of the self-management intervention -CDSMP- on self-efficacy, self-management behaviors and health-related quality of life of women with RA attended in outpatient consultation at a health institution in Bogotá, compared to conventional care.

Specific Objectives. To describe the clinical and sociodemographic variables present in women with RA participating in the study.

To compare the levels of self-efficacy, self-management behaviors, and health-related quality of life of women with RA who received the intervention -CDSMP- before and after its application.

To compare the levels of self-efficacy, self-management and health-related quality of life of women with RA included in the experimental group with the levels of self-efficacy, self-management and health-related quality of life of women with RA in the control group.

Hypothesis

The nursing intervention in self-management CDSMP - is effective in increasing the levels of self-efficacy of women with RA attended in outpatient consultation at a health institution in Bogota compared to conventional care.

The nursing intervention in self-management CDSMP-, is effective in increasing self-management behaviors of women with RA attended in outpatient consultation in a health institution in Bogota compared to conventional care.

The nursing intervention in self-management CDSMP - is effective in increasing the levels of health-related quality of life of women with RA attended in outpatient consultation at a health institution in Bogota compared to conventional care.

ELIGIBILITY:
Inclusion Criteria:

* This study examined women over the age of 18 who were treated at rheumatology outpatient clinics at a health center in Bogotá and had a confirmed diagnosis of rheumatoid arthritis according to the 2010 EULAR/ACR classification criteria.

Exclusion Criteria:

* Women with RA with a comorbid acute process (another or other chronic diseases that the person suffers from and at the time of being identified, are in the exacerbation or crisis phase).
* Women with RA who present cognitive impairment that prevents them from participating in the program or answering the questionnaires due to cognitive impossibility to understand them.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Self-management behaviors | 8 weeks
  For self-management, participants are expected to achieve a high overall score on the self-management behaviors scale, with scores above 80 points.
  The scale consists of 12 items with three dimensions: adherence to treatment (7 items 3, 4, 5, 6, 7, 8 and 12); symptom management (3 items 9, 10 and 11) and knowledge (2 items 1 and 2).
  The answers to the 12 items of the instrument are structured on a scale of 0 to 8 points, the sum of the scores obtained in each item presents the global self-management, the higher the score, the higher the global self-management (0 to 96 points).
  To identify the specific score for each dimension, the sum of the items corresponding to each dimension (knowledge: maximum score 16 points; adherence: 56 points; and symptom management: 24 points) is added together.

SECONDARY OUTCOMES:
Perceived Self-efficacy, | 8 weeks
  For perceived self-efficacy, participants are expected to achieve high overall self-efficacy, with scores of 9 to 10 on the Spanish Arthritis Self-Efficacy-8 scale.
  The scale consists of eight items and two components, the first refers to the possibility of perceiving self-efficacy in reducing pain and performing basic activities of daily living; the second is related to perceived self-efficacy in the control of depressive symptoms due to functional disability resulting from the disease.
  The score for each of the items ranges from 1 to 10, the higher the score the higher the self-efficacy. The total score is the average of the 8 items.
Health-related quality of life | 8 weeks
  In terms of health-related quality of life, participants are expected to achieve high levels of health-related quality of life, with scores of 9 to 10 on the Quality Of Life-Rheumatoid Arthritis Scale-II.
  The scale is composed of eight questions that evaluate different aspects of the quality of life; it is answered by means of a visual numerical scale that goes from one to ten, and then the linear sum of all its components is made and divided by eight, the higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Burbano, Master, Principal Investigator — Universidad Nacional de Colombia; Olga Gómez Ramírez, PhD, Study Director — Universidad Nacional de Colombia; Gerardo Quintana López, Magíster en Epidemiología Clín, Study Chair — Fundación Santa Fe de Bogotá; Ruben Dario Mantilla Hernández, Especialista en Reumatología, Study Chair — Fundación para la Investigación en Dermatología y Reumatología- Funinderma
Locations (1):
- Fundación para la Investigación en Dermatología y Reumatología- Funinderma, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abel WM, DeHaven MJ. An interactive technology enhanced coaching intervention for Black women with hypertension: Randomized controlled trial study protocol. Res Nurs Health. 2021 Feb;44(1):24-36. doi: 10.1002/nur.22090. Epub 2020 Dec 15. PMID 33319386
- [Background] Adepoju OE, Bolin JN, Phillips CD, Zhao H, Ohsfeldt RL, McMaughan DK, Helduser JW, Forjuoh SN. Effects of diabetes self-management programs on time-to-hospitalization among patients with type 2 diabetes: a survival analysis model. Patient Educ Couns. 2014 Apr;95(1):111-7. doi: 10.1016/j.pec.2014.01.001. Epub 2014 Jan 13. PMID 24468198
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Background] Azevedo R, Bernardes M, Fonseca J, Lima A. Smartphone application for rheumatoid arthritis self-management: cross-sectional study revealed the usefulness, willingness to use and patients' needs. Rheumatol Int. 2015 Oct;35(10):1675-85. doi: 10.1007/s00296-015-3270-9. Epub 2015 Apr 24. PMID 25903352
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Barragan-Martinez C, Amaya-Amaya J, Pineda-Tamayo R, Mantilla RD, Castellanos-de la Hoz J, Bernal-Macias S, Rojas-Villarraga A, Anaya JM. Gender differences in Latin-American patients with rheumatoid arthritis. Gend Med. 2012 Dec;9(6):490-510.e5. doi: 10.1016/j.genm.2012.10.005. PMID 23217568
- [Background] Blok AC. A Middle-Range Explanatory Theory of Self-Management Behavior for Collaborative Research and Practice. Nurs Forum. 2017 Apr;52(2):138-146. doi: 10.1111/nuf.12169. Epub 2016 Jul 20. PMID 27438773
- [Background] Cameron-Tucker HL, Wood-Baker R, Owen C, Joseph L, Walters EH. Chronic disease self-management and exercise in COPD as pulmonary rehabilitation: a randomized controlled trial. Int J Chron Obstruct Pulmon Dis. 2014 May 19;9:513-23. doi: 10.2147/COPD.S58478. eCollection 2014. PMID 24876771
- [Background] Cardiel MH. [Present and future of rheumatic diseases in Latin America. Are we prepared to face them?]. Reumatol Clin. 2011 Sep-Oct;7(5):279-80. doi: 10.1016/j.reuma.2010.12.009. Epub 2011 Apr 5. No abstract available. Spanish. PMID 21925442
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krle A-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 Statement: defining standard protocol items for clinical trials. Rev Panam Salud Publica. 2015 Dec;38(6):506-14. PMID 27440100
- [Background] Favalli EG, Biggioggero M, Crotti C, Becciolini A, Raimondo MG, Meroni PL. Sex and Management of Rheumatoid Arthritis. Clin Rev Allergy Immunol. 2019 Jun;56(3):333-345. doi: 10.1007/s12016-018-8672-5. PMID 29372537
- [Background] Forjuoh SN, Bolin JN, Huber JC Jr, Vuong AM, Adepoju OE, Helduser JW, Begaye DS, Robertson A, Moudouni DM, Bonner TJ, McLeroy KR, Ory MG. Behavioral and technological interventions targeting glycemic control in a racially/ethnically diverse population: a randomized controlled trial. BMC Public Health. 2014 Jan 23;14:71. doi: 10.1186/1471-2458-14-71. PMID 24450992
- [Background] Funovits J, Aletaha D, Bykerk V, Combe B, Dougados M, Emery P, Felson D, Hawker G, Hazes JM, Huizinga T, Kay J, Kvien TK, Smolen JS, Symmons D, Tak PP, Silman A. The 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis: methodological report phase I. Ann Rheum Dis. 2010 Sep;69(9):1589-95. doi: 10.1136/ard.2010.130310. PMID 20699242
- [Background] Goeppinger J, Armstrong B, Schwartz T, Ensley D, Brady TJ. Self-management education for persons with arthritis: Managing comorbidity and eliminating health disparities. Arthritis Rheum. 2007 Aug 15;57(6):1081-8. doi: 10.1002/art.22896. PMID 17665471
- [Background] Gonzalez VM, Stewart A, Ritter PL, Lorig K. Translation and validation of arthritis outcome measures into Spanish. Arthritis Rheum. 1995 Oct;38(10):1429-46. doi: 10.1002/art.1780381010. PMID 7575693
- [Background] Grady PA, Gough LL. [Self-management: a comprehensive approach to management of chronic conditions]. Rev Panam Salud Publica. 2015 Mar;37(3):187-94. Spanish. PMID 25988256
- [Background] Griffiths C, Bremner S, Islam K, Sohanpal R, Vidal DL, Dawson C, Foster G, Ramsay J, Feder G, Taylor S, Barnes N, Choudhury A, Packe G, Bayliss E, Trathen D, Moss P, Cook V, Livingstone AE, Eldridge S. Effect of an Education Programme for South Asians with Asthma and Their Clinicians: A Cluster Randomised Controlled Trial (OEDIPUS). PLoS One. 2016 Dec 28;11(12):e0158783. doi: 10.1371/journal.pone.0158783. eCollection 2016. PMID 28030569
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822
- [Background] Home D, Carr M. Rheumatoid arthritis: the role of early intervention and self-management. Br J Community Nurs. 2009 Oct;14(10):432-6. doi: 10.12968/bjcn.2009.14.10.44495. PMID 19966683
- [Background] Iikuni N, Sato E, Hoshi M, Inoue E, Taniguchi A, Hara M, Tomatsu T, Kamatani N, Yamanaka H. The influence of sex on patients with rheumatoid arthritis in a large observational cohort. J Rheumatol. 2009 Mar;36(3):508-11. doi: 10.3899/jrheum.080724. Epub 2009 Feb 4. PMID 19208610
- [Background] Iversen MD, Hammond A, Betteridge N. Self-management of rheumatic diseases: state of the art and future perspectives. Ann Rheum Dis. 2010 Jun;69(6):955-63. doi: 10.1136/ard.2010.129270. Epub 2010 May 6. PMID 20448289
- [Background] Jonker AA, Comijs HC, Knipscheer KC, Deeg DJ. Benefits for elders with vulnerable health from the Chronic Disease Self-management Program (CDSMP) at short and longer term. BMC Geriatr. 2015 Aug 15;15:101. doi: 10.1186/s12877-015-0090-4. PMID 26275714
- [Background] Kneipp SM, Horrell L, Gonzales C, Linnan L, Lee Smith M, Brady T, Trogdon JG. Participation of lower-to-middle wage workers in a study of Chronic Disease Self-Management Program (CDSMP) effectiveness: Implications for reducing chronic disease burden among racial and ethnic minority populations. Public Health Nurs. 2019 Sep;36(5):591-602. doi: 10.1111/phn.12623. Epub 2019 Jun 5. PMID 31168851
- [Background] Lee DM, Weinblatt ME. Rheumatoid arthritis. Lancet. 2001 Sep 15;358(9285):903-11. doi: 10.1016/S0140-6736(01)06075-5. PMID 11567728
- [Background] Lesuis N, Befrits R, Nyberg F, van Vollenhoven RF. Gender and the treatment of immune-mediated chronic inflammatory diseases: rheumatoid arthritis, inflammatory bowel disease and psoriasis: an observational study. BMC Med. 2012 Aug 1;10:82. doi: 10.1186/1741-7015-10-82. PMID 22853635
- [Background] Lin AM, Vickrey BG, Barry F, Lee ML, Ayala-Rivera M, Cheng E, Montoya AV, Mojarro-Huang E, Gomez P, Castro M, Corrales M, Sivers-Teixeira T, Tran JL, Johnson R, Ediss C, Shaby B, Willis P, Sanossian N, Mehta B, Dutta T, Razmara A, Bryg R, Song S, Towfighi A. Factors Associated With Participation in the Chronic Disease Self-Management Program: Findings From the SUCCEED Trial. Stroke. 2020 Oct;51(10):2910-2917. doi: 10.1161/STROKEAHA.119.028022. Epub 2020 Sep 11. PMID 32912091
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lorig K, Laurin J, Holman HR. Arthritis self-management: a study of the effectiveness of patient education for the elderly. Gerontologist. 1984 Oct;24(5):455-7. doi: 10.1093/geront/24.5.455. No abstract available. PMID 6500266
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Lorig K, Ritter PL, Plant K. A disease-specific self-help program compared with a generalized chronic disease self-help program for arthritis patients. Arthritis Rheum. 2005 Dec 15;53(6):950-7. doi: 10.1002/art.21604. PMID 16342084
- [Background] Massardo L, Suarez-Almazor ME, Cardiel MH, Nava A, Levy RA, Laurindo I, Soriano ER, Acevedo-Vazquez E, Millan A, Pineda-Villasenor C, Galarza-Maldonado C, Caballero-Uribe CV, Espinosa-Morales R, Pons-Estel BA. Management of patients with rheumatoid arthritis in Latin America: a consensus position paper from Pan-American League of Associations of Rheumatology and Grupo Latino Americano De Estudio De Artritis Reumatoide. J Clin Rheumatol. 2009 Jun;15(4):203-10. doi: 10.1097/RHU.0b013e3181a90cd8. PMID 19502907
- [Background] Ory MG, Ahn S, Jiang L, Smith ML, Ritter PL, Whitelaw N, Lorig K. Successes of a national study of the Chronic Disease Self-Management Program: meeting the triple aim of health care reform. Med Care. 2013 Nov;51(11):992-8. doi: 10.1097/MLR.0b013e3182a95dd1. PMID 24113813
- [Background] Papakonstantinou D. Work disability and rheumatoid arthritis: Predictive factors. Work. 2021;69(4):1293-1304. doi: 10.3233/WOR-213550. PMID 34366311
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Shigaki CL, Smarr KL, Siva C, Ge B, Musser D, Johnson R. RAHelp: an online intervention for individuals with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1573-81. doi: 10.1002/acr.22042. PMID 23666599
- [Background] Smolen JS, Aletaha D, Bijlsma JW, Breedveld FC, Boumpas D, Burmester G, Combe B, Cutolo M, de Wit M, Dougados M, Emery P, Gibofsky A, Gomez-Reino JJ, Haraoui B, Kalden J, Keystone EC, Kvien TK, McInnes I, Martin-Mola E, Montecucco C, Schoels M, van der Heijde D; T2T Expert Committee. Treating rheumatoid arthritis to target: recommendations of an international task force. Ann Rheum Dis. 2010 Apr;69(4):631-7. doi: 10.1136/ard.2009.123919. Epub 2010 Mar 9. PMID 20215140
- [Background] Tam J, Lacaille D, Liu-Ambrose T, Shaw C, Xie H, Backman CL, Esdaile JM, Miller K, Petrella R, Li LC. Effectiveness of an online self-management tool, OPERAS (an On-demand Program to EmpoweR Active Self-management), for people with rheumatoid arthritis: a research protocol. Trials. 2019 Dec 11;20(1):712. doi: 10.1186/s13063-019-3851-0. PMID 31829286
- [Background] Tengstrand B, Ahlmen M, Hafstrom I. The influence of sex on rheumatoid arthritis: a prospective study of onset and outcome after 2 years. J Rheumatol. 2004 Feb;31(2):214-22. PMID 14760787
- [Background] Theis KA, Helmick CG, Hootman JM. Arthritis burden and impact are greater among U.S. women than men: intervention opportunities. J Womens Health (Larchmt). 2007 May;16(4):441-53. doi: 10.1089/jwh.2007.371. PMID 17521246
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Background] Conn DL, Pan Y, Easley KA, Comeau DL, Carlone JP, Culler SD, Tiliakos A. The effect of the Arthritis Self-Management Program on outcome in African Americans with rheumatoid arthritis served by a public hospital. Clin Rheumatol. 2013 Jan;32(1):49-59. doi: 10.1007/s10067-012-2090-5. Epub 2012 Sep 29. PMID 23053684
- [Background] Twumasi AA, Shao A, Dunlop-Thomas C, Drenkard C, Cooper HLF. Health service utilization among African American women living with systemic lupus erythematosus: perceived impacts of a self-management intervention. Arthritis Res Ther. 2019 Jun 25;21(1):155. doi: 10.1186/s13075-019-1942-7. PMID 31238992
- [Background] Weyand CM, Schmidt D, Wagner U, Goronzy JJ. The influence of sex on the phenotype of rheumatoid arthritis. Arthritis Rheum. 1998 May;41(5):817-22. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-S. PMID 9588732
- [Background] Wilson MG, DeJoy DM, Vandenberg RJ, Padilla HM, Haynes NJ, Zuercher H, Corso P, Lorig K, Smith ML. Translating CDSMP to the Workplace: Results of the Live Healthy Work Healthy Program. Am J Health Promot. 2021 May;35(4):491-502. doi: 10.1177/0890117120968031. Epub 2020 Oct 28. PMID 33111541
- [Background] Wolf TJ, Spiers MJ, Doherty M, Leary EV. The effect of self-management education following mild stroke: an exploratory randomized controlled trial. Top Stroke Rehabil. 2017 Jul;24(5):345-352. doi: 10.1080/10749357.2017.1289687. Epub 2017 Feb 13. PMID 28191861
- [Background] Zuidema R, van Dulmen S, Nijhuis-van der Sanden M, Meek I, van den Ende C, Fransen J, van Gaal B. Efficacy of a Web-Based Self-Management Enhancing Program for Patients with Rheumatoid Arthritis: Explorative Randomized Controlled Trial. J Med Internet Res. 2019 Apr 30;21(4):e12463. doi: 10.2196/12463. PMID 31038461